CLINICAL TRIAL: NCT06518226
Title: Two-Fraction Ultrahypofractionated Radiotherapy With Focal Boost for Intermediate Risk, Localized Prostate Cancer (TURBO): Phase 2, Randomized Controlled Clinical Trial
Brief Title: Two-Fraction Ultrahypofractionated Radiotherapy With Focal Boost for Intermediate Risk, Localized Prostate Cancer
Acronym: TURBO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, J.R.N. van der Voort van Zyp, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL85364.041.23
Record Dates: First submitted 2024-07-05; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Localized Prostate Carcinoma
Keywords: MR-guided adaptive radiotherapy; MRgRT; Quality of life; Patient-reported outcomes; Ultrahypofractionation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrahypofractionated MRgRT in 2 fractions (Experimental): MRgRT to the prostate in 2 fractions of 12 Gy, with a focal boost of 13.5 Gy to the gross tumor volume (GTV), administered over the course of 8 days.
  Interventions: Radiation: Ultrahypofractionated MRgRT in 2 fractions
- Standard of care: MRgRT in 5 fractions (Active Comparator): MRgRT to the prostate in 5 fractions of 7.25 Gy to the prostate without focal boost, administered over the course of 16-18 days.
  Interventions: Radiation: Standard of care: MRgRT in 5 fractions

INTERVENTIONS:
Radiation: Ultrahypofractionated MRgRT in 2 fractions — 2x12 Gy with boost to GTV up to 13.5 Gy
  Arms: Ultrahypofractionated MRgRT in 2 fractions
Radiation: Standard of care: MRgRT in 5 fractions — 5x7.25 Gy
  Arms: Standard of care: MRgRT in 5 fractions

SUMMARY:
The goal of this clinical trial is to assess the non-inferiority irradiating low and intermediate risk, localized prostate cancer in two fractions of radiotherapy, compared to five fractions of radiotherapy which is the standard of care. The main question it aims to answer are:

- Do participants in the interventional arm have more physician-reported grade 2 or higher acute Common Terminology Criteria for Adverse Events (CTCAE) genitourinary (GU) side effects?

Participants in the intervention arm will receive two fractions of radiotherapy, in which the prostate is irradiated with 12 Gy per fraction and the tumor receives a boost of up to 13.5 Gray (Gy), over the course of 8 days. Those in the control arm will receive five fractions of radiotherapy of 7.25 Gy each to the prostate, without a boost to the tumor, over the course of 16-18 days.

DETAILED DESCRIPTION:
Rationale: Hypofractionation in prostate cancer radiotherapy has already led to a drastic reduction in fractionation scheme from 35 fractions to the now standard 5 fractions for patients with intermediate risk prostate cancer. Currently, biochemical progression free survival is at approximately 90% at five-year follow-up for intermediate risk prostate cancer patients, which leaves little to no room for further improvement in oncological outcomes. However, with an ageing population and a subsequently higher volume of patients with localized prostate cancer, there is a need to improve and optimize current treatment options. Treatment cost within the field of prostate oncology will further increase over the years to come, and an early economic health evaluation has demonstrated that a 2-fractionation scheme with MRI-guided radiotherapy (MRgRT) for intermediate risk prostate cancer patients is cost effective compared to the standard of care 5 fractions scheme.

Previous research demonstrated the feasibility of delivering high doses of radiation in only two fractions, both in silico as well as in a clinical setting using a conventional CT-guided linear accelerator. With the introduction of MRgRT, however, it has become possible to deliver higher doses of radiation with more accuracy, while limiting genitourinary (GU) and gastrointestinal (GI) toxicity. This leads us to believe that improvements can be made both in terms of costs as well as patient reported quality of life.

Objective: To assess the effectiveness, safety and feasibility of treating patients with localized, intermediate risk prostate cancer who will receive radiation therapy in two fractions of 12 Gy with a boost to the gross tumor volume of 13.5 Gy per fraction in 8 days, as compared to standard care (36.25 Gy in five fractions in 16-18 days), on an ELEKTA Unity MR-Linac system.

Study design: Single-center, prospective, open label, phase II randomized controlled trial.

Study population: Men with localized, intermediate risk prostate cancer who are to receive radiation therapy with curative intent. Exclusion criteria are previous radical prostatectomy, presence of contraindications for MRI or conditions which predispose to increased morbidity and/or toxicity (such as colitis ulcerosa, Crohn's disease), previous pelvic radiotherapy, metal pelvic implants causing artefact of MR-imaging, and previous invasive malignancy within the last 5 year (excluding cutaneous basal cell carcinoma)

Intervention: Participants in the intervention arm will receive two fractions of 12 Gy to the clinical target volume (CTV) with a boost up to 13.5 Gy to the gross tumor volume (GTV) of radiation in a time span of 8 days on an MR-linac. Those in the control arm will receive five fractions of 7.25 Gy in a time span of 16-18 days on an MR-linac, as per standard care.

Main study parameters/endpoints: Difference in proportion of participants with acute CTCAE grade 2 or higher GU toxicity.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This trial will be nested in the observational Multiple OutcoMe EvaluatioN of radiation Therapy Using the MR-Linac (MOMENTUM) study, and participants will receive QOL questionnaires which are already embedded within this cohort. Therefore, participants are not subjected to an additional burden during the course and follow-up period of this study. In a recently published study, there was no evidence that hypofractionation caused more GU and/or GI grade ≥2 toxicity. Radiobiologically, the low alpha/beta ratio of prostate cancer makes it more sensitive to higher doses of radiation in fewer fractions, which is in fact the essence of the ultrahypofractionation scheme that we offer in the interventional arm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histopathological confirmation of prostate adenocarcinoma requiring radical treatment
* European Association of Urology (EAU) intermediate risk prostate cancer, defined as Prostate Specific Antigen (PSA) level of < 20 ng/ml, Gleason score ≤ 7, cT1c-cT2b/iT3a (non-bulky, < 20mm)
* Written informed consent
* Ability and willingness to comply with Patient Reported Outcome Measure (PROM) questionnaires schedule throughout the study
* Inclusion in the Multi-OutcoMe EvaluatioN of radiation Therapy Using the MR-Linac Study (MOMENTUM)

Exclusion Criteria:

* Contraindications to MRI
* International Prostate Symptom Score (IPSS) of 15 or higher
* Prostate volume > 80 cc
* Comorbidities which predispose to significant toxicity (e.g., inflammatory bowel disease)
* Metal pelvic implants which cause artefact on MR-imaging sequences
* Previous radical prostatectomy
* Previous pelvic radiotherapy
* Previous invasive malignancy within the last 5 years, excluding basal cell carcinoma of the skin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute grade >= 2 genitourinary (GU) physician-reported toxicity | 90 days after treatment
  This is scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 scale. Scores will be retrieved from the hospital information system.

SECONDARY OUTCOMES:
Incidence of acute grade >= 2 gastrointestinal (GI) physician-reported toxicity | Up to 5 years
  This is scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 scale. Scores will be retrieved from the hospital information system.
Incidences of late grade >= 2 GU physician-reported toxicity | Up to 5 years
  This is scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 scale. Scores will be retrieved from the hospital information system.
Incidences of acute grade >= 2 GI physician-reported toxicity | Up to 5 years
  This is scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 scale. Scores will be retrieved from the hospital information system.
Oncological treatment related quality of life (QoL) | Up to 5 years
  Oncological treatment related quality of life is captured through the generic European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire(QLQ)-C30. It includes 5 functional scales (physical, role, emotional, cognitive and social), three symptom scales, a global health scale, and six single items. All of these scales and items measures range in score from 0 to 100. A high score on functional or global health status scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Patient reported Health related quality of life (HRQoL) | Up to 5 years
  Generic patient reported quality of life is captured by the EuroQol (EQ)-5D-5L questionnaire. This includes a descriptive system questionnaire and visual analogue scale (VAS). The descriptive system scores five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) from 1 to 5 where 1 means having no problems, and 5 means extreme problems or unable to participate. The digits can be combined in a 5-digit code to describe the overall health status. For example, 12111. The VAS records the overall current health on a vertical visual analogue scale from 0 to 100, respectively 'the worst health you can imagine' to 'the best health you can imagine'.
Patient reported prostate cancer-specific quality of life (QoL). | Up to 5 years
  Prostate cancer-specific patient reported quality of life is captured by the tumor specific European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire(QLQ)-C30. The questionnaire consists of functional and symptom scales. All of these scales and items measures range in score from 0 to 100. A high score on functional scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Biochemical progression free survival (bPFS) | Up to 5 years
  Prostate Specific Antigen (PSA) levels in ng/mL will be retrieved from the hospital information system. Biochemical recurrence is defined as serum PSA levels that are 2 ng/mL higher than the nadir PSA achieved after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Westley RL, Biscombe K, Dunlop A, Mitchell A, Oelfke U, Nill S, Murray J, Pathmanathan A, Hafeez S, Parker C, Ratnakumaran R, Alexander S, Herbert T, Hall E, Tree AC. Interim Toxicity Analysis From the Randomized HERMES Trial of 2- and 5-Fraction Magnetic Resonance Imaging-Guided Adaptive Prostate Radiation Therapy. Int J Radiat Oncol Biol Phys. 2024 Mar 1;118(3):682-687. doi: 10.1016/j.ijrobp.2023.09.032. Epub 2023 Sep 29. PMID 37776979
- [Derived] Lalmahomed TA, Monninkhof EM, van Rijssel MJ, van Melick HHE, Verkooijen HM, de Boer JCJ, van der Voort van Zyp JRN. Two-fraction Ultrahypofractionated Radiotherapy with focal BOost for intermediate-risk, localized prostate cancer (TURBO): study protocol of a phase II, randomized controlled clinical trial. Trials. 2025 Dec 29;26(1):586. doi: 10.1186/s13063-025-09297-5. PMID 41466435